CLINICAL TRIAL: NCT04606212
Title: Losartan Effects on the Emotion Processing in Humans
Brief Title: The Effects of Losartan on Emotion Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-73
Record Dates: First submitted 2020-10-09; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: Losartan; emotion processing
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental)
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Losartan — administration of losartan (50 mg) (oral)
  Arms: Losartan group
Drug: Placebo Oral Tablet — administration of placebo (oral)
  Arms: Placebo group

SUMMARY:
The aim of the study is to investigate the effect of losartan (50mg, single dose) on salience processing

DETAILED DESCRIPTION:
In a double-blind, between-subject, placebo-controlled design the effects of a single dose of losartan (50mg) on salience processing in healthy participants will be examined. The study will adopt a previously validated visual Oddball fMRI paradigm, starting 90 minutes after subjects receive 50mg losartan or placebo. The task requires participants to respond to emotional and novelty oddballs. Neural activity will be assessed by the acquisition of functional magnetic resonance imaging (fMRI) data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury
* medical or psychiatric illness
* hypertension

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Neural activity as measured by BOLD fMRI during processing of emotional and novel stimuli | 105 to 145 minutes after treatment administration
  During the oddball paradigm a series of pictures will be presented in rapid succession. Some of the stimuli are oddballs, with respect to emotional content (highly threatening stimuli) or novelty (novel stimuli). Neural activity will be measured by functional magnetic resonance imaging (fMRI). The fMRI data will be examined using a Generalized Linear Model approach. The analysis will examine neural activity in terms of the blood oxygenation dependent (BOLD) response towards threatening and novel oddballs. Effects of treatment on the BOLD response towards threatening and novel oddballs will be examined by comparing the losartan- and placebo-treated subjects.

SECONDARY OUTCOMES:
Neural activity as measured by BOLD fMRI during processing of different categories of emotional and novel stimuli | 105 to 145 minutes after treatment administration
  The oddball paradigm will include different stimulus categories (animal pictures and human faces). Each category will include oddballs, with respect to emotional content (highly threatening stimuli) or novelty (novel stimuli). Neural activity will be measured by functional magnetic resonance imaging (fMRI). The fMRI data will be examined using a Generalized Linear Model approach. The analysis will examine neural activity differences between the stimulus categories (animal pictures, human face pictures) in terms of the blood oxygenation dependent (BOLD) response. Effects of treatment on the BOLD response towards different stimulus categories will be examined by comparing the losartan- and placebo-treated subjects.
Accuracy for target oddballs | 105 to 145 minutes after treatment administration
  Before the paradigm two stimuli will be designated as 'target' and subjects are required to respond by button press to this target. The accuracy for target detection will be computed. Effects of treatment will be examined by comparing the losartan- and placebo-treated subjects.
Reaction times for target oddballs | 105 to 145 minutes after treatment administration
  Before the paradigm two stimuli will be designated as 'target' and subjects are required to respond by button press to this target. The reaction times for correctly identified targets will be computed. Effects of treatment will be examined by comparing reaction times between the losartan- and placebo-treated subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No